CLINICAL TRIAL: NCT06000397
Title: Parents' Enhanced Reminder Intervention to Improve Children's Timely Completion of Immunization Series of Pneumococcal Vaccine at the 12-month's Visit
Brief Title: Reminder Emails to Improve Pneumococcal Vaccine Completion at 12 Months of Age
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20220678-01H
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Pneumococcal Vaccines; Immunization Coverage
Keywords: Vaccine coverage; Vaccine uptake

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced reminders (Experimental)
  Interventions: Other: Enhanced reminders
- Standard notifications (Active Comparator)
  Interventions: Other: Standard CANImmunize notifications

INTERVENTIONS:
Other: Enhanced reminders — The intervention is sending enhanced (modality and frequency) of reminders to CANImmunize App users, in addition to the standard notifications. Specifically:
  * Deliver reminders and recall emails to parents or guardians of infants waiting for their 12-month dose of pneumococcal vaccine,
  * Add additional information about the benefits, safety and effectiveness of the pneumococcal vaccine to support increased uptake, and
  * Provide tips to improve parents' or guardians' self-efficacy in circumventing barriers to timely immunization of children at the 12-month's visit
  Arms: Enhanced reminders
Other: Standard CANImmunize notifications — Push notifications at two time points:
  * two weeks prior to the immunization due date
  * one week after the immunization due date
  Arms: Standard notifications

SUMMARY:
The goal of this clinical trial is to assess the effectiveness of enhanced email reminders in improving vaccine coverage at the 12-month visit in CANImmunize app users. The main questions it aims to answer are:

* Do enhanced email reminders improve coverage of the 12- month dose of the pneumococcal vaccine and the timely completion of its immunization series at the 12-month's visit in CANImmunize app users?
* What are the predictors of predictors of timely completion of the 12-month's series of pneumococcal vaccines in the CANImmunize app users?

Participants will be randomized to either receive enhanced reminder/recall materials via email or the standard CANImmunize notifications. Researchers will compare the enhanced reminder group to the standard notification group to see if there is a difference in vaccine coverage at the 12-month visit.

ELIGIBILITY:
Inclusion Criteria

To be included in the study, CANImmunize account holders must have:

* Enabled the reception to receive emails from CANImmunize, and
* Record(s) for an infant aged between 10- and 11-months, who have already received the earlier doses of the pneumococcal vaccine in accordance with their provincial/territorial routine immunization schedule.

Exclusion Criteria

* The account holder (parent, or guardian of the child) has an inactive or undelivered email address, or
* No record(s) for an infant aged 10- and 11-months, or
* The record for the 10- or 11-month-old indicates that he/she has not received the prior pneumococcal vaccine doses.

Ages: 10 Months to 11 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 700 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Receipt of 12-month pneumococcal vaccine | 12 months of age
  Receipt of the 12-month dose of the pneumococcal vaccine as recorded in the CANImmunize immunization record

SECONDARY OUTCOMES:
Timeliness of 12-month pneumococcal vaccine | 12-13 months of age will be considered as timely, after 13 months considered late
  Age at receipt of the 12-month dose of the pneumococcal vaccine as recorded in the CANImmunize immunization record

CONTACTS AND LOCATIONS:
Locations (1):
- CANImmunize, Ottawa, Canada